CLINICAL TRIAL: NCT05500898
Title: A Phase I Clinical Trial to Evaluate the Safety and Drug Interactions Between DWP16001 and in Combination With DWC202204 and DWC202205 in Healthy Adult Volunteers
Brief Title: Drug-Drug Interaction of DWP16001 in Combination With DWC202204 and DWC202205 in Healthy Male Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001108
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental)
  Interventions: Drug: DWP16001
- Experimental 2 (Experimental)
  Interventions: Drug: DWC202204+DWC202205
- Experimental 3 (Experimental)
  Interventions: Drug: DWP16001+DWC202204+DWC202205

INTERVENTIONS:
Drug: DWP16001 — Tablets, Oral, multiple doses of DWP16001
  Arms: Experimental 1
Drug: DWC202204+DWC202205 — Tablets, Oral, multiple doses of DWC202204 and DWC202205 in combination
  Arms: Experimental 2
Drug: DWP16001+DWC202204+DWC202205 — Tablets, Oral, DWP16001 , multiple doses of DWC202204 and DWC202205 in combination
  Arms: Experimental 3

SUMMARY:
The purpose of this study is to evaluate drug-drug interaction by comparing the pharmacokinetics (PK)/pharmacodynamics (PD), safety, and tolerability of single/multiple doses of DWP16001 , DWC202204 and DWC202205 alone or in combination in healthy male adults.

DETAILED DESCRIPTION:
* Open label, multiple dose, 2 part, two period, single sequence design. This study is conducted on open label because it evaluates PK/PD parameters that are not affected by the blind. Volunteers who are suitable for the inclusion criteria are granted the final target number before the first dosage, receiving a fixed IP, and conducting a planned clinical trial schedule.

After having a rest period (7 days) in which the drug received is sufficiently metabolized and lost, the IP of the next period is administered.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults ≥ 19 years of age at the time of the screening procedure
2. 18.5 ≤ body mass index (BMI) ≤ 27.0
3. Voluntarily decided to participate in the study and provided written consent prior to the screening procedure after receiving a detailed explanation on this study and fully understanding the information
4. Is eligible to participate in the study at the discretion of the investigator by a physical examination, laboratory test, and medical history questionnaire, etc.

Exclusion Criteria:

1. Presence or prior history of a clinically significant hepatic, renal, nervous, respiratory, endocrine, hematologic and oncologic, cardiovascular, urogenital, psychiatric disorder
2. Presence or prior history of a gastrointestinal disorder (e.g., gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc.), or prior history of gastrointestinal surgery (except for simple appendectomy or hernia surgery) that may affect the safety and PK/PD assessment of the study drug.
3. Hypersensitivity to, or history of clinically significant hypersensitivity to drugs including DWP16001 and other drugs of the same class (SGLT2 inhibitors), drugs including gemigliptin and other drugs of the same class, metformin and other drugs (aspirin, antibiotics, etc.)
4. Considered ineligible for the study by the investigator for reasons including laboratory test results

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-08-26 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss of DWP16001 | [Time Frame: 0-72 hours]
  Peak Plasma Concetration at steady-state
AUCtau,ss of DWP16001 | [Time Frame: 0-72 hours]
  Area under the plasma concentration versus time curve at Tau, steady-state
Cmax,ss of DWC202204 and DWC202205 | [Time Frame: 0-24 hours]
  Peak Plasma Concetration at steady-state
AUCtau,ss of DWC202204 and DWC202205 | [Time Frame: 0-24 hours]
  Area under the plasma concentration versus time curve at Tau, steady-state